CLINICAL TRIAL: NCT05574270
Title: Clinical Investigation of a Small Aperture Extended Depth of Focus Intraocular Lens in Patients With Complex Corneas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC8-204-EXP2
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cataract; Presbyopia; Irregular Astigmatism
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IC-8 IOL Group (Experimental): A monofocal or monofocal toric IOL implanted in the first eye of a subject and the IC-8 IOL implanted in the second eye.
  Interventions: Device: IC-8 Intraocular Lens (IOL)

INTERVENTIONS:
Device: IC-8 Intraocular Lens (IOL) — A small aperture extended depth of focus hydrophobic acrylic intraocular lens.
  Other Names: IC-8 IOL

SUMMARY:
The objective of this study is to evaluate the clinical outcomes of the IC-8 IOL implanted in patients with complex corneas after crystalline lens removal.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, non-randomized, single-arm clinical investigation with planned postoperative follow-up of 4-6 months. The monocular and binocular performance of the subjects will be evaluated.

The objective of this study is to evaluate the clinical outcomes of the IC-8 IOL implanted in patients with complex corneas after crystalline lens removal.

The co-primary effectiveness endpoints are monocular uncorrected distance, intermediate, and near visual acuities at 4-6 Months postoperative. The primary safety endpoint is best-corrected distance visual acuity at 4-6 Months postoperative. The secondary safety endpoint is photopic and mesopic contrast sensitivity at 4-6 Months postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 22 years of age;
2. Able to comprehend and have signed a statement of informed consent;
3. Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visit(s);
4. Planned crystalline lens removal by phacoemulsification, with or without femtosecond laser-assisted extraction, and posterior chamber IOL implantation;
5. Planned cataract removal or planned clear lens exchange in both eyes
6. Potential for postoperative best-corrected distance visual acuity (BCDVA) of 20/32 or better after crystalline lens removal;
7. Having complex corneas with irregular astigmatism
8. Having clear central cornea
9. Having best-corrected distance visual acuity (BCDVA) or 20/40 or worse in either eye with or without a glare source (patients with bilateral cataract).

Exclusion Criteria:

1. Requiring an IC-8 IOL outside the available spherical power range;
2. Pharmacologically dilated pupil size less than 6 mm in either eye;
3. Preoperative corneal astigmatism >1.50 diopters in the eye to be implanted with the IC-8 IOL;
4. Active or recurrent anterior segment pathology;
5. Presence of ocular abnormalities or conditions (other than corneal irregularities) as specified by the protocol;
6. Congenital bilateral cataracts;
7. Previous ocular surgery as specified by the protocol;
8. Conditions requiring planned ocular surgical intervention;
9. Severe dry eye or other conditions (such as hormonal fluctuations) that could lead to unstable refraction and/or visual acuity measurements or eye discomfort even with ocular lubricants or dry eye medication;
10. Use of systemic or ocular medications as specified by the protocol;
11. Concurrent participation or participation in any clinical investigation up to 30 days prior to preoperative visit;
12. Patient is pregnant or nursing.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Monocular uncorrected distance visual acuity (UCDVA) | 4-6 Months
  Mean acuity from the IC-8 IOL eye at 4-6 Months is statistically better compared to preoperative
Monocular uncorrected intermediate visual acuity (UCIVA) | 4-6 Months
  Mean acuity from the IC-8 IOL eye at 4-6 Months is statistically better compared to preoperative
Monocular uncorrected near visual acuity (UCNVA) | 4-6 Months
  Mean acuity from the IC-8 IOL eye at 4-6 Months is statistically better compared to preoperative
Monocular best-corrected distance visual acuity (BCDVA) in the IC-8 IOL eye | 4-6 Months
  Mean best-corrected distance visual acuity (BCDVA) in the IC-8 IOL eye at 4-6 Months is not statistically worse than 0.2 logMAR

SECONDARY OUTCOMES:
Monocular and Binocular Contrast Sensitivity | 4-6 Months
  Photopic and Mesopic contrast sensitivity (with and without glare) in each eye and both eyes will be analyzed. No success criterion or hypothesis testing.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Michna, Ph.D., Study Director — AcuFocus, Inc.
Locations (2):
- Asian Eye Institute, Makati City, Philippines
- Singapore National Eye Centre (SNEC); Singapore Eye Research Institute (SERI), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No